CLINICAL TRIAL: NCT01168141
Title: Assessment of the Effects of the Specific Endothelin-A Antagonist ZD4054 on Prostate Cancer Biomarkers in Patients With Castrate-resistant Metastatic Disease
Brief Title: Window Study of ZD4054 in Metastatic Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Ms Angela Ball, Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 08_CLPHA_54
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-06

CONDITIONS: Prostate Cancer; Metastasis
Keywords: Castrate-resistant prostate cancer with bone metastasis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ZD4054 — 10mg ZD4054 daily in tablet form
  Other Names: Zibotentan

SUMMARY:
This is a prospective study in which patients with castrate-resistant prostate cancer and bone metastases will undergo imaging, donate blood, bone marrow and urine samples, and where possible primary tumour and bone metastatic tissue, before and during treatment with ZD4054, an orally active specific endothelin-A antagonist. The samples will be used primarily for biomarker studies, and it is hypothesized that these will inform on the mechanism of action of this drug. Magnetic Resonance Imaging (MRI) will be performed to evaluate emerging functional imaging endpoints as markers of early response in bone metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmation of prostate adenocarcinoma
* documented evidence of bone metastasis on bone scan or MRI
* biochemical progression of prostate cancer
* surgically or medically castrate with serum testosterone ≤2.4nmol/L
* ECOG performance status 0 - 2
* life expectancy of 6 months or more.

Exclusion Criteria:

* radiotherapy to bone lesion or prostatic bed within 4 weeks of starting study treatment.
* prior targeted cancer therapies (such as gefitinib, bevacizumab)
* systemic radionuclide therapy within 12 weeks of starting study treatment.
* current therapy, within 4 weeks of study entry with potent inhibitors of CYP3A4 (ketoconazole, itraconazole, ritonavir, indinavir, erythromycin, troleandomycin, clarithromycin, diltiazem and verapamil), inhibitors of CYPs 2D6 and 2C9 (quinidine and fluconazole), and potent P450 inducers (phenytoin, rifampicin, carbamazepine and phenobarbitone)
* definite or suspected personal history or family history of adverse drug reactions, or hypersensitivity to drugs that are endothelin antagonists
* ineligibility for MRI scanning includes standard MRI criteria (for example, metal implants such as cochlear implants, cardiac pacemakers, heart valves, aneurysm clips and metal fragments in eyes) and patients known to be allergic to gadolinium-based MRI contrast agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Changes in tissue biomarkers | 6 weeks
Changes in blood-borne biomarkers | 12 weeks
Changes in imaging biomarkers | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom